CLINICAL TRIAL: NCT06101771
Title: Assessment of Epicardial Fat Thickness in Children With Familial Dyslipidemia in Assiut University Children Hospital, Egypt
Brief Title: Assessment of Epicardial Fat Thickness in Children With Familial Dyslipidemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Mamdouh Wahib Tadros, Resident doctor of Pediatrics, Faculty of Medicine, Assiut University, Principal Investigator., Assiut University
Other Study IDs: children with dyslipidemia
Record Dates: First submitted 2023-09-19; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dyslipidemia: Normal weight children more than 1 month and till age of 18 years that attend Assiut University children Hospital with Clinical manifestation:
  1. Non-symptomatic accidentally discovered dyslipidemia.
  2. Steatorrhea.
  3. Fatty liver.
  Interventions: Diagnostic Test: echoCARDIOGRAPHY

INTERVENTIONS:
Diagnostic Test: echoCARDIOGRAPHY — Assessment of epicardial fat thickness in children with familial dyslipidemia

SUMMARY:
Aim of the study: 1- Detect common types of familial dyslipidemia. 2- Significance and relationship between Epicardial fat thickness and familial dyslipidemia.

DETAILED DESCRIPTION:
Dyslipidemias or dyslipoproteinemias are quantitative changes in total cholesterol concentration, respective fractions, or triglycerides in the plasma. Lipids, such as cholesterol or triglycerides, are absorbed from the intestines and are carried throughout the body via lipoproteins for energy, steroid production, or bile acid formation . Major contributors to these pathways are cholesterol, low-density lipoprotein cholesterol (LDL-C), triglycerides, and high-density lipoprotein (HDL). An imbalance of any of these factors, either from organic or nonorganic causes, can lead to dyslipidemia. Dyslipidemias can result from primary lipoprotein metabolism changes due to different genetic causes (primary dyslipidemias) or as a consequence of exogenous factors or other pathologies (secondary dyslipidemias). Primary dyslipidemia can be due to familial disorders as well. Autosomal dominant mutations cause most cases of familial hypercholesterolemia in LDL receptors, which causes an elevation in LDL-C levels. Other mutations in the cholesterol pathway have been identified but are less common. Several health behaviors can have effects and increase lipid levels. Examples include tobacco use, physical inactivity, nutrition, and obesity. Specifically, nutrition risk factors include the insufficient consumption of fruits, nuts/seeds, vegetables, or high consumption of saturated fats.

The heart and vessels are surrounded by layers of adipose tissue, which is a complex organ composed of adipocytes, stromal cells, macrophages, and a neuronal network, all nourished by a rich microcirculation . The layers of adipose tissue surrounding the heart can be subdivided into intra- and extrapericardial fat. Their thicknesses and volumes can be quantified by echocardiography and CT or magnetic resonance imaging, respectively.

The term extrapericardial fat defines thoracic adipose tissue external to the parietal pericardium. It originates from primitive thoracic mesenchymal cells and thus derives its blood supply from noncoronary sources. Intrapericardial fat is further subdivided into epicardial and pericardial fat. Anatomically, Epicardial and pericardial adipose tissues are clearly different.

Epicardial fat is located between the outer wall of the myocardium and the visceral layer of pericardium. Epicardial adipose tissue (EAT) is a component of visceral adiposity and mediates cardiac function and atherosclerosis via expression of several bioactive molecules.

EAT is a measure of the adipose tissue between the myocardium and visceral pericardium which can be visualized using transthoracic echocardiogram as a non-invasive assessment of EAT. Some studies have used EAT as a marker for metabolic syndrome; however, it does not have standard utility related to other cardiac syndromes. This fat layer buffers the coronary arteries from cardiac contraction and arterial pulse wave while providing the myocardium with necessary substrate through diffusion of free fatty acids. 4 When there is a surplus of energy, free fatty acids are readily converted into triglycerides and stored in epicardial adipocytes, increasing the volume of the epicardial adipose layer and serving as a triglyceride depot for the myocardium to draw from during periods of higher energy needs. Studies in adults suggest that increased EAT results in greater cytokine production in the fat directly surrounding the coronary vessels, including tumor necrosis factor-αas well as several interleukins. These cytokines contribute to atherosclerosis by increasing lipolysis, increasing inflammation, and causing endothelial dysfunction. Endothelial dysfunction coupled with migration of macrophages, basophils, and other cells further exacerbate plaque formation and eventually causes disruption in the structure of the intima and flow within the lumen.8,9Recent studies suggest that increased EAT is predictive of incident CVD in adults with T1D independent of traditional CVD risk factors such as BMI. Although the majority of studies examining EAT have been conducted in the adult population, EAT has been measured in pediatric studies of obesity and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight children more than 1 month and till age of 18 years that attend Assiut University children Hospital with Clinical manifestation:

  1. Non-symptomatic accidentally discovered dyslipidemia.
  2. Steatorrhea.
  3. Fatty liver

Exclusion Criteria:

1- Patients who had poor echo window : chest deformities, chronic lung disease, pericardial and/or pleural effusion on transthoracic echocardiography, and chronic kidney disease were not included in the study.

2. Congenital heart diseases. 3. Children with liver diseases that cause 2ry dyslipidemia. 4. Children with Diabetes that cause 2ry dyslipidemia

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Setting: Tertiary care center ( Assiut University children Hospital) (AUCH) from Sep 2023 to Sep 2025.
  Normal weight children more than 1 month and till age of 18 years that attend Assiut University children Hospital with Clinical manifestation:
  1. Non-symptomatic accidentally discovered dyslipidemia.
  2. Steatorrhea.
  3. Fatty liver.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
assessment epicardial fat thickness in children with familial dyslipidemia | baseline
  All cases included in the study will be evaluated by:
  1. - Fasting lipid profile: Total cholesterol, High-density lipoprotein (HDL) cholesterol, Low-density lipoprotein (LDL) cholesterol, Triglycerides (TG). (18)
  2. - Transthoracic Echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Mohamed Kotb, Lecturer of Pediatrics, Study Director — Assiut University; Mohamed Abou Bakr Sobeih, Lecturer of Pediatrics, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided